CLINICAL TRIAL: NCT04777097
Title: Does Preeclampsia Affect Blood Loss During a Caesarean Procedure
Brief Title: Blood Loss and Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00123
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Pre-Eclampsia; Complicating Pregnancy; Blood Loss; Coagulation Disorder
Keywords: Pre-eclampsia; blood-loss; impaired coagulation
MeSH Terms: conditions — Pre-Eclampsia; Pregnancy Complications; Hemorrhage; Hemostatic Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy pregnant women: Healthy patients who receive a cesarean operation
  Interventions: Other: Blood sample
- Pre-eclampsia: Patients with pre-eclampsia who receive a caesarean operation
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Two blood sample will be drawn. On the day of operation and the first postoperative day.

SUMMARY:
Study of blood loss in preeclamptic patients using mathematical formulae

DETAILED DESCRIPTION:
Pre-eclampsia is a symptom complex that occurs in 2-5% of all pregnancies and leads to significant morbidity and mortality. It is associated with a risk of impaired coagulation caused by a reduced platelet count, very rarely by disseminated intravascular coagulation disorders. The degree of clotting correlates with the severity of preeclampsia. It is planned to calculate the blood loss using mathematical formulas and to compare the different blood loss in the two groups (preeclampsia vs. healthy pregnant women). Furthermore, this project will try to correlate the blood loss with the underlying coagulation situation. The aim is to be able to better assess the bleeding risk in healthy pregnant women, but also in pre-eclamptic patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Elective or urgent caesarean section
* Written informed consent

Exclusion Criteria:

* Emergency caesarean section
* Familial coagulation disorder
* Hematological disorders that affect the platelet count, e.g. myelodysplastic syndrome (MDS)
* Taking anticoagulants
* Taking aspirin in the last 14 days
* Use of NSARs in the last 24 hours

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Patients with pre-eclampsia planed for cesarean section vs. healty pregnant women, planmned for cesarean section
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Blood-Loss | day 1
  Corelation between blood loss and coagulation parameters will be calculated

SECONDARY OUTCOMES:
Coagulation parameter | day 1
  Impact of pre-eclampsia on the coagulation parameters

CONTACTS AND LOCATIONS:
Overall Officials: Marco P Zalunardo, Principal Investigator — Institut of Anesthesiology University Hospital Zurich
Locations (1):
- University Hospital Zurich, Institute for Anesthesiology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Brecher ME, Monk T, Goodnough LT. A standardized method for calculating blood loss. Transfusion. 1997 Oct;37(10):1070-4. doi: 10.1046/j.1537-2995.1997.371098016448.x. PMID 9354828
- [Result] Theusinger OM, Kind SL, Seifert B, Borgeat L, Gerber C, Spahn DR. Patient blood management in orthopaedic surgery: a four-year follow-up of transfusion requirements and blood loss from 2008 to 2011 at the Balgrist University Hospital in Zurich, Switzerland. Blood Transfus. 2014 Apr;12(2):195-203. doi: 10.2450/2014.0306-13. PMID 24931841
- [Result] de Lange NM, Lance MD, de Groot R, Beckers EA, Henskens YM, Scheepers HC. Obstetric hemorrhage and coagulation: an update. Thromboelastography, thromboelastometry, and conventional coagulation tests in the diagnosis and prediction of postpartum hemorrhage. Obstet Gynecol Surv. 2012 Jul;67(7):426-35. doi: 10.1097/OGX.0b013e3182605861. PMID 22926249